CLINICAL TRIAL: NCT02515006
Title: Randomized Controlled Trial of Homeopathy Compared With Treatment As Usual for Persistent Insomnia in Patients With Cancer
Brief Title: Impact of Homeopathy for Persistent Insomnia in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adwin Life Care (Industry)
Collaborators: Center For Homeopathy Research, India (Unknown); Sonal Foundation, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Adwin/chr/1121
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Insomnia; Cancer
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Homeopathy (Experimental): Individualized homeopathy treatment as a supportive care
  Interventions: Other: Homeopathy Medicine
- Control (No Intervention): Usual Care

INTERVENTIONS:
Other: Homeopathy Medicine — Homeopathy, or homeopathic medicine, is a holistic system of treatment. Individualized homeopathy remedy was based on the most characteristic and clear mental symptoms. Secondly, general symptoms were taken into account.C-potencies were provided and manufactured according to the Homeopathic Pharmacopoeia and Hahnemann's methodology. Each individualized homeopathic remedy were be prescribed in C-potencies
  Arms: Homeopathy

SUMMARY:
Persistent insomnia is highly prevalent complaint in cancer survivors, but is seldom satisfactorily addressed. The adaptation to cancer care of a validated, cost-effective intervention may offer a practicable solution. The aim of this study was to investigate the clinical effectiveness of homeopathy for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to begin chemotherapy or radiotherapy
* chemotherapy or radiotherapy
* meet diagnostic criteria for chronic insomnia (i.e., lasting for at least one month)
* Chronic insomnia has been defined in previous research:as the presence of (1) three or more episodes of insomnia (i.e., ≥ 30minuteSOL, ≥ 60minute wake after sleep onset (WASO), or ≤ 6.5 hour total sleep time (TST) per night) of per week and (2) daytime effects of insomnia, such as irritability, difficulty concentrating, or fatigue for at least one month.
* have the permission of their oncologists to participate.

Exclusion Criteria:

* untreated alcohol or substance abuse or dependence,
* bipolar, or psychotic disordermedical conditions such as seizure disorder, restless leg disorder, or Parkinson's disease
* untreated sleep disorders such as sleep apnea
* Taking other alternative medicines

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in sleep efficiency on the Insomnia Severity Index | From baseline to 6 Months

SECONDARY OUTCOMES:
Change in Anxiety and Depression on Hospital Anxiety Depression Scale | From Baseline to 6 Months
Change in Quality of Life on Short Form-36 Scale | From Baseline to 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Tejendra H Patel, BBA, Study Director — Center for Homeopathy Research; Neha Sharma, PhD, Principal Investigator — NMP Medical Research Institute; Govind Sharma, MD, Study Chair — Adwin Life Care
Locations (2):
- India (2):
  - Center for Homeopathy Research, Ahmedabad, Gujarat
  - Center for Homeopathy Research, Jaipur, Rajasthan